CLINICAL TRIAL: NCT00836407
Title: A Phase Ib Trial Evaluating the Safety and Feasibility of Ipilimumab (BMS-734016) Alone or in Combination With Allogeneic Pancreatic Tumor Cells Transfected With a GM-CSF Gene for the Treatment of Locally Advanced, Unresectable or Metastatic Pancreatic Adenocarcinoma
Brief Title: Ipilimumab +/- Vaccine Therapy in Treating Patients With Locally Advanced, Unresectable or Metastatic Pancreatic Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: J0834; BMS # CA184-081
Record Dates: First submitted 2009-02-03; First posted 2009-02-04 (Estimated); Results first posted 2013-12-10 (Estimated); Last update posted 2020-02-24 (Actual); Status verified 2020-02

CONDITIONS: Pancreatic Cancer
Keywords: pancreatic cancer; vaccine; immunotherapy; antibody; CTLA-4
MeSH Terms: conditions — Pancreatic Neoplasms; Diabetes Mellitus, Insulin-Dependent, 12 | interventions — Ipilimumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm 1: Ipilimumab Alone (Experimental): Ipilimumab alone
  Interventions: Drug: Ipilimumab
- Arm 2: Ipilimumab + Pancreatic Cancer Vaccine (Experimental): Ipilimumab + Pancreatic Cancer Vaccine
  Interventions: Drug: Ipilimumab; Biological: Pancreatic Cancer Vaccine

INTERVENTIONS:
Drug: Ipilimumab — Ipilimumab (10mg/kg) will be administered intravenously at weeks 1, 4, 7 and 10. Subjects will also be offered maintenance phase dosing every 12 weeks.
  Other Names: BMS-734016; MDX-010
Biological: Pancreatic Cancer Vaccine — The Pancreatic Cancer Vaccine (5E8 cells) will be administered intradermally at weeks 1, 4, 7 and 10. Subjects will also be offered maintenance phase dosing every 12 weeks.
  Other Names: PANC 10.05 pcDNA-1/GM-Neo and PANC 6.03 pcDNA-1 neo vaccine
  Arms: Arm 2: Ipilimumab + Pancreatic Cancer Vaccine

SUMMARY:
Research Hypothesis: Ipilimumab (an antibody that blocks negative signals to T cells) administered alone or in combination with a pancreatic cancer vaccine (allogeneic pancreatic tumor cells transfected with a GM-CSF gene), has an acceptable safety profile in subjects with locally advanced, unresectable or metastatic pancreatic adenocarcinoma.

Primary Objective: To determine the safety profile of ipilimumab alone or in combination with a pancreatic cancer vaccine in subjects with locally advanced, unresectable or metastatic pancreatic adenocarcinoma.

Secondary Objectives:

* To estimate overall survival (OS) which will serve as the primary efficacy signal.
* To explore an association of T cell responses and immunological responses with OS in patients receiving treatment.
* To estimate overall response rate (ORR), immune related best overall response rate (irBOR), progression free survival (PFS), and duration of response in patients receiving treatment.
* To explore an association between immune-related adverse events (IRAEs) and ORR.
* To measure tumor marker kinetics (CA 19-9) in patients receiving treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Documented cancer of the pancreas who have failed (or are not candidates for) standard therapy
2. ECOG Performance Status of 0 to 1
3. Adequate organ function as defined by study-specified laboratory tests
4. Must use acceptable form of birth control through the study and for 28 days after final dose of study drug
5. Signed informed consent form
6. Willing and able to comply with study procedures

Exclusion Criteria:

1. Currently have or have history of certain study-specified heart, liver, kidney, lung, neurological, immune or other medical conditions
2. Clinical metabolic or laboratory abnormalities defined as Grade 3 or 4 of the National Cancer Institute's (NCI's) Common Terminology Criteria for Adverse Events (CTCAE), version 3.0
3. Systemically active steroids
4. Another investigational product within 28 days prior to receiving study drug
5. Major surgery or significant traumatic injury (or unhealed surgical wounds) occurring within 28 days prior to receiving study drug
6. Infection with HIV, hepatitis B or C at screening
7. Pregnant or lactating
8. Conditions, including alcohol or drug dependence, or intercurrent illness that would affect the patient's ability to comply with study visits and procedures

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2009-02; Primary Completion 2012-07 (Actual); Study Completion 2012-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dung Le, MD, Principal Investigator — The Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins
Locations (1):
- Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins, Baltimore, Maryland, United States

REFERENCES:
- [Result] Le DT, Lutz E, Uram JN, Sugar EA, Onners B, Solt S, Zheng L, Diaz LA Jr, Donehower RC, Jaffee EM, Laheru DA. Evaluation of ipilimumab in combination with allogeneic pancreatic tumor cells transfected with a GM-CSF gene in previously treated pancreatic cancer. J Immunother. 2013 Sep;36(7):382-9. doi: 10.1097/CJI.0b013e31829fb7a2. PMID 23924790
- [Derived] Hopkins AC, Yarchoan M, Durham JN, Yusko EC, Rytlewski JA, Robins HS, Laheru DA, Le DT, Lutz ER, Jaffee EM. T cell receptor repertoire features associated with survival in immunotherapy-treated pancreatic ductal adenocarcinoma. JCI Insight. 2018 Jul 12;3(13):e122092. doi: 10.1172/jci.insight.122092. PMID 29997287

RESULTS

PARTICIPANT FLOW:
Groups:
- Arm 1: Ipilimumab Alone: Ipilimumab (10mg/kg) will be administered intravenously at weeks 1, 4, 7 and 10. Subjects will also be offered maintenance phase dosing every 12 weeks.
- Arm 2: Ipilimumab + Pancreatic Cancer Vaccine: Drug: Ipilimumab Ipilimumab (10mg/kg) will be administered intravenously at weeks 1, 4, 7 and 10. Subjects will also be offered maintenance phase dosing every 12 weeks.
  Biological/Vaccine: Pancreatic Cancer Vaccine The Pancreatic Cancer Vaccine (5E8 cells) will be administered intradermally at weeks 1, 4, 7 and 10. Subjects will also be offered maintenance phase dosing every 12 weeks.
Period: Overall Study
Arm/Group | Arm 1: Ipilimumab Alone | Arm 2: Ipilimumab + Pancreatic Cancer Vaccine
Started | 15 | 15
Completed | 4 | 7
Not Completed | 11 | 8

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm 1: Ipilimumab Alone | Arm 2: Ipilimumab + Pancreatic Cancer Vaccine | Total
Number analyzed (Participants) | 15 | 15 | 30
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 9 | 10 | 19
  >=65 years | 6 | 5 | 11
Age, Continuous [Mean (Standard Deviation); unit: years] | 62.3 (7.8) | 61.9 (8.9) | 62.1 (8.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 5 | 9
  Male | 11 | 10 | 21
Region of Enrollment [Number; unit: participants]
  United States | 15 | 15 | 30

OUTCOME MEASURES:

1. Primary Outcome: Percent of Patients Experiencing an Unacceptable Toxicity
Description: Unacceptable toxicity is defined as drug related >grade 4 AEs or grade 3 AEs including IRAEs not improving to < grade 2 under therapy within 2 weeks. In addition, > grade 2 eye pain or reduction of visual acuity that does not respond to topical therapy and does not improve to < grade 1 severity within 2 weeks of starting therapy, or requires systemic therapy is an unacceptable toxicity.
Time Frame: 4 years
Measure: Number; unit: Percentage of Participants
Arm/Group | Arm 1: Ipilimumab Alone | Arm 2: Ipilimumab + Pancreatic Cancer Vaccine
Number analyzed (Participants) | 15 | 15
Percentage of Participants | 6.67 | 6.67

2. Secondary Outcome: Overall Survival (OS)
Description: OS will be measured from date of randomization until death or end of follow-up (OS will be censored on the date the subject was last known to be alive for subjects without documentation of death at the time of analysis).
Time Frame: 4 years
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Arm 1: Ipilimumab Alone | Arm 2: Ipilimumab + Pancreatic Cancer Vaccine
Number analyzed (Participants) | 15 | 15
Months | 3.6 [2.5 to 9.2] | 5.7 [4.3 to 14.7]

3. Secondary Outcome: Overall Response Rate (ORR)
Description: ORR is defined as the number of patients achieving a complete response (CR) or partial response (PR) based on the Response Evaluation Criteria in Solid Tumors (RECIST 1.1) during the first 6 months of treatment. CR = disappearance of all target lesions, PR is =>30% decrease in sum of diameters of target lesions, progressive disease (PD) is >20% increase in sum of diameters of target lesions, stable disease (SD) is <30% decrease or <20% increase in sum of diameters of target lesions. Estimation based on the Kaplan-Meier curve.
Time Frame: 6 months
Reporting Status: Not Posted

4. Secondary Outcome: Immune Related Best Overall Response Rate (irBOR)
Description: Immune Related Best Overall Response (BOR) is the best response recorded from the start of the study treatment until the disease progression/recurrence based on the Response Evaluation Criteria in Solid Tumors (RECIST 1.1). Estimation based on the Kaplan-Meier curve.
Time Frame: 4 years
Reporting Status: Not Posted

5. Secondary Outcome: Progression Free Survival (PFS)
Description: PFS is defined as the number of months from the date of randomization to disease progression (progressive disease [PD] or relapse from complete response [CR] as assessed using RECIST 1.1 criteria) or death due to any cause. Per RECIST 1.1 criteria, CR = disappearance of all target lesions, Partial Response (PR) is =>30% decrease in sum of diameters of target lesions, Progressive Disease (PD) is >20% increase in sum of diameters of target lesions, Stable Disease (SD) is <30% decrease or <20% increase in sum of diameters of target lesions.
Time Frame: 6 months
Reporting Status: Not Posted

ADVERSE EVENTS:
Arm/Group | Arm 1: Ipilimumab Alone | Arm 2: Ipilimumab + Pancreatic Cancer Vaccine
Serious Adverse Events (participants affected / at risk) | 3/15 | 1/15
Other Adverse Events (participants affected / at risk) | 11/15 | 15/15
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm 1: Ipilimumab Alone (N=15) | Arm 2: Ipilimumab + Pancreatic Cancer Vaccine (N=15)
Nephritis (Renal and urinary disorders) | 1 (1) | 0 (0)
Colitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Guillain-Barre Syndrome (Nervous system disorders) | 1 (1) | 0 (0)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | Arm 1: Ipilimumab Alone (N=15) | Arm 2: Ipilimumab + Pancreatic Cancer Vaccine (N=15)
Adrenal insufficiency (Endocrine disorders) | 0 (0) | 1 (1)
Hypophysitis (Endocrine disorders) | 2 (2) | 1 (1)
Conjuntivitis (Eye disorders) | 1 (1) | 0 (0)
Colitis (Gastrointestinal disorders) | 2 (2) | 4 (4)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Anorexia (Gastrointestinal disorders) | 0 (0) | 2 (3)
Cramps (Gastrointestinal disorders) | 1 (1) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 0 (0) | 2 (2)
Dry eye (Eye disorders) | 1 (1) | 0 (0)
Dry skin (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Fatigue (General disorders) | 0 (0) | 6 (7)
Fever (General disorders) | 3 (5) | 5 (12)
Flu-like symptoms (General disorders) | 2 (2) | 4 (8)
Headache (Nervous system disorders) | 0 (0) | 3 (6)
Nausea (Gastrointestinal disorders) | 1 (1) | 2 (2)
Pruritis (Skin and subcutaneous tissue disorders) | 4 (5) | 6 (14)
Rash (Skin and subcutaneous tissue disorders) | 6 (7) | 9 (23)
Urticaria (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
Blister, vaccine site (Skin and subcutaneous tissue disorders) | 0/0 (0) | 2 (9)
Hyperpigmentation, vaccine site (Skin and subcutaneous tissue disorders) | 0/0 (0) | 1 (1)
Pruritis, vaccine site (Skin and subcutaneous tissue disorders) | 0/0 (0) | 14 (40)
Erythema, vaccine site (Skin and subcutaneous tissue disorders) | 0/0 (0) | 15 (48)
Induration, vaccine site (Skin and subcutaneous tissue disorders) | 0/0 (0) | 15 (53)
Tenderness, vaccine site (Skin and subcutaneous tissue disorders) | 0/0 (0) | 13 (33)
Urticaria, vaccine site (Skin and subcutaneous tissue disorders) | 0/0 (0) | 1 (1)
Vaccine Site Flare (Skin and subcutaneous tissue disorders) | 0/0 (0) | 1 (11)
Warmth, vaccine site (Skin and subcutaneous tissue disorders) | 0/0 (0) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No